CLINICAL TRIAL: NCT05045833
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Multiple Ascending Dose Study to Assess the Pharmacokinetics, Safety, and Tolerability of Orally Administered SYN 020 Delayed Release Capsules in Healthy Subjects
Brief Title: Multiple Ascending Dose Study to Assess the Pharmacokinetics, Safety, and Tolerability of Orally Administered SYN 020
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theriva Biologics, Inc. (Industry)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: SB-1-020-002
Record Dates: First submitted 2021-09-09; First posted 2021-09-16 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2021-09

CONDITIONS: Enteritis Caused by Radiation

STUDY DESIGN:
Intervention Model Description: Multiple Ascending Dose Escalation
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blinded Investigational Drug (Active and Placebo)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 5 mg SYN-020 (Experimental): 1 x 5 mg oral capsule, 14 days, dosing every 12 hours, 6 subjects receive active, 2 subjects receive placebo
  Interventions: Drug: SYN-020 Delayed Release Capsule
- 15 mg SYN-020 (Experimental): 1 x 15 mg oral capsule, 14 days, dosing every 12 hours, 6 subjects receive active, 2 subjects receive placebo
  Interventions: Drug: SYN-020 Delayed Release Capsule
- 45 mg SYN-020 (Experimental): 3 x 15 mg oral capsules, 14 days, dosing every 12 hours, 6 subjects receive active, 2 subjects receive placebo
  Interventions: Drug: SYN-020 Delayed Release Capsule
- 75 mg SYN-020 (Experimental): 5 x 15 mg oral capsules, 14 days, dosing every 12 hours, 6 subjects receive active, 2 subjects receive placebo
  Interventions: Drug: SYN-020 Delayed Release Capsule
- ≤ 75 mg SYN-020 (new formulation) (Experimental): ≤ 5 x 15 mg oral capsules, 14 days, dosing every 12 hours, 6 subjects receive active, 2 subjects receive placebo
  Interventions: Drug: SYN-020 Delayed Release Capsule

INTERVENTIONS:
Drug: SYN-020 Delayed Release Capsule — Oral administration (by mouth)

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, multiple-ascending-dose study to assess the PK, safety, and tolerability of SYN-020 oral delayed release capsules (SYN 020) in healthy adults. At least 1 exploratory PD endpoint will also be assessed.

DETAILED DESCRIPTION:
Randomization to treatment will be stratified by sex, with equal numbers of males and females receiving each treatment in each cohort. Up to 5 ascending-dose cohorts of 8 subjects each will be enrolled, and all cohorts will be conducted as planned or until the safety data do not support further escalation. SYN-020 (or placebo) will be administered every 12 hours for 14 consecutive days at escalating doses of 5, 15, 45, and 75 mg in Cohorts 1 through 4, and at a dose not to exceed 75 mg in Cohort 5.

Subjects will be screened within 28 days before admission to the clinical research unit (CRU). For each cohort, eligible subjects will be admitted to the CRU on Day -1, and subjects who remain eligible will receive the first dose of study drug in the morning (AM) of Day 1. Subjects will receive study drug every 12 hours for 14 consecutive days. No restriction in food or fluids is required around dosing for any dose other than the AM dose on Days 1 and 14. Subjects will also fast overnight before blood samples are collected for clinical laboratory and/or PD tests on Days 2, 6, 8, 10, 14, and at the follow-up visit on Day 35. A standard Western diet appropriate for a Phase 1 study will be provided at approximately the same times each day during confinement, with each cohort receiving the same meals.

Subjects will be discharged from the CRU after the End of Study (EOS) procedures are completed in the AM on Day 15 and will return to the CRU for a follow-up visit on Day 35.

For PK assessment, blood samples (primarily on Days 1 and 14) and feces (pre-dose and over selected 48 hour time intervals) will be collected for analysis of SYN 020 concentrations.

For PD assessment, blood will be collected and analyzed (or stored for future analysis) for at least 1 of the exploratory endpoints. Fecal samples for PD assessment will be taken from the feces collected for PK assessment. These investigations will explore potential biomarkers for future SYN 020 indications and will be strictly and directly related to the pharmacology of SYN 020. While gastrointestinal microbiome/metabolome analyses include genotyping of the gut bacteria, no human genotyping will be performed.

Safety and tolerability will be monitored throughout the study. Safety assessments will include clinical laboratory tests, vital signs, 12-lead ECGs, physical examinations, monitoring for AEs, and ADA testing. Adverse event data will be collected from the time of informed consent through the follow-up visit at Day 35 or until the AE resolves or becomes stable.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to read, write, and comprehend English at a sufficient level to understand study-related materials, has provided written informed consent before any study-related procedure was performed, and is willing and able to comply with all testing and study requirements.
2. Subject is a healthy male or female, at least 18 years of age.
3. Subject does not use any tobacco or nicotine product (for example, cigarette, pipe, e cigarette, vape, smokeless tobacco) and has not used any tobacco or nicotine product for at least 2 months before CRU admission.
4. Subject has a BMI of 18.5 to <35 kg/m2. Note: Approximately 50% of subjects should have BMI > 25 kg/m2; however, randomization is not based on BMI.
5. Subject is healthy based on physical examination, clinical laboratory tests, 12-lead ECG, and vital signs.
6. Subject is willing to minimize the risk of inducing pregnancy from the time of signing the ICF to at least either 90 days (males) or 30 days (females) after the last study drug dose by following the procedures below.

   If male: Must agree to abstain from donating sperm for at least 90 days after the study drug dose.

   If male has a female sexual partner of childbearing potential: He must ALSO agree to use at least one of the following medically acceptable methods of contraception for at least 90 days after the study drug dose:
   * Bilateral vasectomy performed at least 1 year before screening
   * Use of a condom or diaphragm plus either contraceptive sponge, foam, or jelly
   * Complete abstinence from heterosexual intercourse; periodic abstinence is not acceptable

   If a sexually active female of childbearing potential (defined as a female after puberty who is not postmenopausal for at least 1 year or surgically sterile): Must agree to use at least one of the following medically acceptable methods of contraception for at least 30 days after the study drug dose:
   * Intrauterine device (hormonal or non-hormonal, inserted 2 or more cycles before Screening)
   * Hormonal contraception (stable use for 2 or more cycles before Screening) administered orally or by depot injection or implant, transdermal system, or vaginal ring
   * Bilateral tubal ligation
   * Male partner with a bilateral vasectomy performed at least 1 year before screening
   * Barrier contraception: Use of a condom or diaphragm plus either contraceptive sponge, foam, or jelly
   * Complete abstinence from heterosexual intercourse; periodic abstinence is not acceptable
7. If female, subject has a negative serum pregnancy test at Screening and upon CRU admission.
8. Subject usually has at least 1 bowel movement a day based on self-reporting.

Exclusion Criteria:

1. Subject has a history or the presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, vascular, metabolic, collagen, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
2. Subject has any known malabsorption syndrome or history of gastrointestinal surgery that could compromise the study objectives.
3. Subject has used any medication (prescription or non-prescription) or herbal supplement other than prescription hormone replacement therapy (eg, thyroid, testosterone, estrogen) within 21 days before CRU admission or, if female, has used hormonal contraception if use has not been stable for 2 or more cycles before Screening.
4. Subject is pregnant, breastfeeding, or not using a medically accepted method of contraception.
5. Subject is unable to abstain from artificial sweeteners (eg, aspartame, acesulfame potassium, advantame, saccharin, stevia, and sucralose) from CRU admission to CRU discharge.
6. Subject has a positive urine drug or alcohol test at Screening or CRU admission OR has a history of drug/alcohol abuse within 12 months before Screening.
7. Subject has donated more than 500 mL blood during the 3-month period before CRU admission.
8. Subject has known intolerance of study drug or ingredients.
9. In the judgment of the Investigator, subject has any factor (eg, other treatment) that could invalidate the study result.
10. Subject is currently enrolled in another clinical study or has received an investigational drug or device within 30 days or within a time period consistent with a washout period of 5 half-lives before signing the ICF, whichever is longer.
11. Subject has already participated in this or a previous SYN 020 study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
SYN-020 systemic absorption | Day 1 to Day 15
  Analysis of SYN-020 level present in blood
SYN-020 presence in feces | Day -1 to Day 14
  Analysis of SYN-020 level present in feces

SECONDARY OUTCOMES:
Monitoring for Safety and Tolerability | Day 1 to Day 35
  Adverse Events, CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Clinical Research LLC, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No